CLINICAL TRIAL: NCT03791515
Title: Clinical Characteristics and Pathophysiology of Post-Traumatic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Associate Professor of Neurology, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-18011477
Record Dates: First submitted 2018-07-27; First posted 2019-01-02 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2018-12

CONDITIONS: Post-Traumatic Headache; Concussion, Mild
MeSH Terms: conditions — Post-Traumatic Headache; Brain Concussion | interventions — Calcitonin Gene-Related Peptide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 100 patients with PPTH and 100 healthy controls will undergo a deep phenotyping of clinical characteristics and associated comorbidities. This is followed by a single MRI-session for all subjects.
  Lastly, the 30 patients with PPTH will participate in a randomized, double-blind, placebo-controlled, 2-way crossover study. These patients will be allocated to receive intravenous infusion of CGRP or placebo (isotonic saline) over 20 minutes on 2 study days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcitonin Gene-Related Peptide (CGRP) (Active Comparator): 30 patients with PPTH will be allocated to receive intravenous infusion of 1.5 µg/min calcitonin-gene related peptide over 20 minutes
  Other Name: CGRP
  Interventions: Drug: Calcitonin Gene-Related Peptide
- Placebo (Placebo Comparator): 30 patients with PPTH wil be allocated to receive 40 mL Placebo (isotonic saline) over 20 minutes.
  Other Name: Isotonic Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin Gene-Related Peptide — A randomized clinical trial with a double-blinded, randomized, placebo-controlled crossover design. 30 PPTH patients will be included. All participants will receive continuous intravenous infusion of 1.5 µg/min CGRP over 20 min.
  The following variables will be recorded before, during and after infusion (every 10 min over 60 min): headache intensity on a verbal rating scale from 0 to 10 and headache characteristics. At 90 min, participants will be discharged and instructed to fill out a headache diary for 24 hours from start of infusion.
  Other Names: CGRP
  Arms: Calcitonin Gene-Related Peptide (CGRP)
Drug: Placebo — A randomized clinical trial with a double-blinded, randomized, placebo-controlled crossover design. 30 PPTH patients will be included. All participants will receive continuous intravenous infusion of 40 mL placebo (isotonic saline) over 20 min.
  The following variables will be recorded before, during and after infusion (every 10 min over 60 min): headache intensity on a verbal rating scale from 0 to 10 and headache characteristics. At 90 min, participants will be discharged and instructed to fill out a headache diary for 24 hours from start of infusion.
  Other Names: Isotonic Saline
  Arms: Placebo

SUMMARY:
To better understand the clinical characteristics and complex pathophysiological events that constitute persistent post-traumatic headache (PPTH) and to identify possible calcitonin gene-related peptide (CGRP) hypersensitivity in PPTH patients.

DETAILED DESCRIPTION:
The present project will embark upon identifying novel PTH-specific biomarkers by incorporating a plethora of scientific approaches. First, clinical biomarkers will be assessed by deep phenotyping of clinical characteristics and associated comorbidities using a semi-structured interview and multiple validated questionnaires. Second, biochemical biomarkers will be determined by plasma levels measurements of blood markers for headache hypersensitivity and neuronal/axonal damage. Third, imaging biomarkers will be established by magnetic resonance imaging (MRI) to assess structural and functional changes in the brain. Lastly, molecular biomarkers will be identified by examining whether intravenous infusion of calcitonin gene-related peptide (CGRP) provokes headache attacks mimicking the usual headache phenotype in subjects with PTH. This would determine whether PTH patients exhibit hypersensitivity to CGRP (molecular biomarker) and advance our understanding of the complex pathophysiological events that constitute the headache phenotypes in PTH sufferers.

ELIGIBILITY:
Inclusion Criteria for PPTH patients:

* 18-65 years of age
* Subject has PPTH in accordance with the diagnostic criteria of the International Headache Society (IHS)
* Concussion (mild traumatic brain injury) occured > 12 months ago
* Subject, who are fertile women, must be on safe contraceptives

Exclusion Criteria for PPTH patients:

* Pre-trauma existing primary headache disorder (maximum 1 day/per month with tension-type headache) and medication-overuse headache
* > 1 episode with a sustained concussion
* Whiplash
* Pregnant or lactating women
* Cardiovascular disease of any kind
* Hypertension on the experimental day
* Hypotension on the experimental day
* Pre-trauma existing psychiatric disorder of any kind - unless well-regulated
* Any anamnestic or clinical signs of any kind deemed relevant for the study by the physician examining the subject
* Any MRI contraindication and a wish of not being informed about unexpected MRI changes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Headache Characteristics | 50 minutes
  Headache characteristics will be assessed using a semi-structured interview.
Headache Characteristics | 10 minutes
  Headache characteristics will be assessed using Headache Under-Response to Treatment Index (HURT-Index) questionnaire. The total score ranges from 0 to 24 with a higher score indicating a lower effectiveness of intervention against headache.
Cognitive Function | 10 minutes
  Cognitive function will be assessed using Montreal Cognitive Assessment (MoCA) questionnaire. The total score ranges from 0 to 30 points. The MoCA is divided into 7 subscores: visuospatial/executive (5 points); naming (3 points); memory (5 points for delayed recall); attention (6 points); language (3 points); abstraction (2 points); and orientation (6 points). One point is added if the subject has ≤12 years of education. A total of 30 points may be given. A score ≤25 indicates some degree of cognitive impairment.
Depression | 10 minutes
  Depression will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. The total score ranges from 0-21.
  A score of 0-7 points is regarded as being in the normal range. A score of 8-10 points is suggestive of a depressive state (borderline abnormal).
  A score of 11-21 points indicates a probable presence of a depressive state (abnormal).
Anxiety | 10 minutes
  Anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire.
  The total score ranges from 0-21. A score of 0-7 points is regarded as being in the normal range. A score of 8-10 points is suggestive of a state of anxiety (borderline abnormal).
  A score of 11-21 points indicates a probable presence of an anxiety disorder (abnormal).
Allodynia | 10 minutes
  Allodynia will be assessed using Allodynia Symptom Checklist (ASC-12) questionnaire. The total score ranges from 0-24 points.
  A score of 0-2 suggests no allodynia. A score of 3-5 suggests mild allodynia. A score of 6-8 suggests moderate allodynia. A score of 9 or more suggests severe allodynia.
Post-Traumatic Stress Disorder | 10 minutes
  Post-traumatic stress disorder will be assessed using Harvard Trauma Questionnaire (HTQ). The total score ranges from 16-64. The total score is divided with 16 and a clinical cut-off score of 2.5 is set to be indicative of PTSD.
Quality of Sleep: Pittsburgh Sleep Quality Index (PSQ-I) | 10 minutes
  Quality of Sleep will be assessed using Pittsburgh Sleep Quality Index (PSQ-I). The measure consists of 19 individual items, creating 7 components that produce one global score. The total PSQ-I score ranges from 0 to 21 with lower scores indicating a healthier sleep quality.
Muscle Tenderness | 10 minutes
  Muscle tenderness will be assessed using Total Tenderness Score (TTS). The total score ranges from 0-48 with higher scores indicating a higher degree of muscle tenderness.
Pressure Pain Threshold | 10 minutes
  Pressure Pain Threshold will be assessed using an Algometer.
Cortical Density | 10 minutes
  Cortical density will be assessed using Voxel-Based Morphometry.
Cortical Thickness | 10 minutes
  Cortical thickness will be assessed using Surface-Based Morphometry
Number and Location of Microhemorrhages | 6 minutes
  The number and location of microhemorrhages will be assessed using Susceptibility-Weighted Imaging.
White Matter Structural Fiber Integrity | 10 minutes
  The white matter structural fiber integrity will be assessed using Diffusion Tensor Imaging
Number and Location of White Matter Lesions | 6 minutes
  The number and location of white matter lesions will be assessed using T2-weighted Fluid-Attenuated Inversion Recovery.
Cerebral Blood Flow | 7 minutes
  Cerebral blood flow will be assessed using arterial spin labelling (ASL).
Brain Network Functional Connectivity | 11 minutes
  Brain network functional connectivity will be assessed using blood oxygen level-dependent functional magnetic resonance imaging.
Incidence of Headache Exacerbation with Migraine-Like Features | 60 minutes
  Migraine-like features are defined as headache fulfilling at least two of the following four characteristics:
  1. Unilateral location
  2. Pulsating quality
  3. Moderate or severe pain intensity
  4. Aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs)
  And during headache at least one of the following must be fulfilled:
  1. Nausea and/or vomiting
  2. Photophobia and phonophobia
  3. Headache mimicking the usual exacerbated headache with migraine-like features
  If the participant fulfills these criteria at baseline, then incidence of exacerbated headache with migraine-like features is defined as:
  - An increase in headache intensity combined with an increase in the degree nausea and/or photophobia and phonophobia (based on a mild / moderate / severe scale)
Headache Area under the Curve | 12 hours
  Headache area under the curve is defined as headache intensity x duration up to 12 h after CGRP infusion
Time to Maximum Headache | 12 hours
  Time to maximum headache score on CGRP day compared to placebo day will be assessed using a headache questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schytz, MD, Principal Investigator — Associate Professor
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schytz HW, Smilkov E, Carroll I, Dobrocky T, Al-Khazali HM, Tolnai D, Jensen RH, Amin FM. No evidence of intracranial hypotension in persistent post-traumatic headache: A magnetic resonance imaging study. Cephalalgia. 2025 Apr;45(4):3331024251325556. doi: 10.1177/03331024251325556. Epub 2025 Apr 21. PMID 40255022